CLINICAL TRIAL: NCT01507207
Title: Pediatric Dysphagia Outcomes After Injection Laryngoplasty for Type I Laryngeal Cleft
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Maria de Lourdes Quintanilla-Dieck, MD, Resident Physician, Department of Otolaryngology Head & Neck Surgery, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 7850
Record Dates: First submitted 2012-01-04; First posted 2012-01-10 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Dysphagia; Aspiration; Quality of Life
Keywords: Dysphagia; aspiration; pediatric; injection laryngoplasty
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Injection laryngoplasty — Patients will undergo a direct microlaryngoscopy in the operating room for diagnostic purposes. In patients in whom laryngeal cleft is diagnosed, injection laryngoplasty will be carried out using sodium carboxymethylcellulose aqueous gel (commercial name Radiesse) injection material.

SUMMARY:
Type I laryngeal cleft evaluation and treatment in the pediatric population is an emerging science. The largest published series of pediatric patients with type I laryngeal clefts shows conflicting evidence in terms of outcomes, resolution of dysphagia and method of treatment. A comparison of quality of life outcomes before and after injection laryngoplasty has not been carried out. The investigators hypothesize that injection laryngoplasty significantly improves symptoms and quality of life related to dysphagia in a pediatric population with laryngeal clefts.

DETAILED DESCRIPTION:
Dysphagia with aspiration is a common disorder in the pediatric population. Aspiration with feeds is diagnosed on modified barium swallow studies and patients are referred to the pediatric otolaryngologist to assess the airway for a possible laryngeal cleft. Type I laryngeal cleft can lead to dysphagia and aspiration in young children. However, diagnosis of type I laryngeal cleft can be difficult and subjective at microlaryngoscopy in the operating room. Type I laryngeal cleft evaluation and treatment in the pediatric population is an emerging science. The largest published series of pediatric patients with type I laryngeal clefts shows conflicting evidence in terms of outcomes, resolution of dysphagia and method of treatment. It is generally recommended to do an injection laryngoplasty at the time of airway evaluation as a diagnostic and therapeutic measure. Improvement in symptoms supports the diagnosis and can serve as either definitive treatment with repeated injections or as a preemptive treatment in preparation for surgical repair. A comparison of quality of life outcomes before and after injection laryngoplasty has not been carried out. Thus, the aim of this study is to determine if injection laryngoplasty improves symptoms and quality of life related to dysphagia in a pediatric population with laryngeal clefts.

ELIGIBILITY:
Inclusion Criteria:

* chief complaint of dysphagia and/or aspiration detected on a clinical swallow assessment and/or modified barium swallow study
* able to withstand general anesthesia and direct microlaryngoscopy in the operating room

Exclusion Criteria:

* inability or parent refusal to undergo procedure under general anesthesia in the operating room

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2015-05-15 (Actual); Study Completion 2015-05-15 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | 3-4 months after procedure
  Measured via previously validated pediatric quality of life survey for dysphagia

CONTACTS AND LOCATIONS:
Overall Officials: Carol MacArthur, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University - Doernbecher Children's Hospital, Portland, Oregon, United States

REFERENCES:
- [Background] Cohen MS, Zhuang L, Simons JP, Chi DH, Maguire RC, Mehta DK. Injection laryngoplasty for type 1 laryngeal cleft in children. Otolaryngol Head Neck Surg. 2011 May;144(5):789-93. doi: 10.1177/0194599810395082. PMID 21493369
- [Background] Clayburgh D, Milczuk H, Gorsek S, Sinden N, Bowman K, MacArthur C. Efficacy of tonsillectomy for pediatric patients with Dysphagia and tonsillar hypertrophy. Arch Otolaryngol Head Neck Surg. 2011 Dec;137(12):1197-202. doi: 10.1001/archoto.2011.196. PMID 22183897